

# √ CathVision

AUTOMATED ASSESSMENT OF PULMONARY VEIN ISOLATION USING A NOVEL EP RECORDING SYSTEM (PVISION)

# **Statistical Analysis Plan**

30 Aug 2022

#### **SPONSOR**

CathVision ApS
Titangade 11
DK-2200
Copenhagen, DENMARK

#### **CRO**

AKRN Scientific Consulting S.L.





#### **Table of Contents** 1.0 ACRONYMS AND ABBREVIATIONS......5 2.0 SYNOPSIS OF STUDY DESIGN ......7 3.0 3.1 Purpose of Statistical Analysis Plan ......7 3.2 Clinical Investigation Objectives.......7 3.3 Clinical Investigation Design ......7 3.4 3.4.1 3.4.2 Safety endpoint.......8 3.4.3 Secondary performance endpoints ......8 3.5 Randomization and blinding.....8 ANALYSIS CONSIDERATIONS......9 4.0 4.1 Analysis Populations ......9 4.1.1 Intent-to-treat population (ITT) ......9 4.1.2 Per-protocol treatment (PPT)......9 4.2 4.3 4.3.1 4.3.2 4.4 4.4.1 4.4.2 4.4.3 4.5 4.6 4.7 4.8 4.9 4.10 4.11 4.12 5.0 DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA......15 5.1 5.2 5.3 5.4





| 5.5 | Number of Subject Imbalance | . 15 |
|-----|-----------------------------|------|
| 6.0 | | |
| 7.0 | APPENDICES | . 17 |





# 1.0 ACRONYMS AND ABBREVIATIONS

| Term | Definition |
|---|---|
| AE | Adverse Event |
| ADE | Adverse Device Effect |
| ВРМ | Beats-Per-Minute |
| CDF | Cumulative Distribution Function |
| CIP | Clinical Investigation Plan |
| CI | Confidence Interval |
| d | Superiority limit |
| EP | Electrophysiology |
| EGM | Electrogram |
| FN | False Negative |
| FP | False Positive |
| ITT | Intent-To-Treat |
| NSR | Non-Sinus Rhythm |
| RF | Radiofrequency |
| р | Proportion |
| PFA | Pulsed-field ablation |
| PPT | Per-Protocol-Treatment |
| PV | Pulmonary Vein |
| PVI | Pulmonary Vein Isolation |
| SAE | Serious Adverse Event |
| SADE | Serious Adverse Device Effect |
| SD | Standard Deviation |
| SE | Sensitivity: Is the ability of a test/procedure to correctly identify those with the disease (true positive rate) |
| SP | Specificity: Is the ability of the test to correctly identify those without the disease (true negative rate). |
| SR | Sinus Rhythm |
| TN | True Negative |
| TP | True Positive |
| UADE | Unanticipated Adverse Device Effect |
| USADE | Unanticipated Serious Adverse Device Effect |



# 2.0 APPLICABLE DOCUMENTS

| External references | | | |
|---|---|---|---|
| Document Type | Document<br>Number | Document Name | Version |
| ISO Standard<br>14155:2020 | N/A | ISO 14155:2020 — Clinical investigation of medical devices for human subjects — Good clinical practice | 2020 |
| ICH E9 | N/A | Statistical Principles for Clinical Trials | 01-SEP-1998 |
| EU Regulation | N/A | Regulation (EU) 2017/745 | N/A |
| Internal references | | | |
| Study Protocol | CPVI-002 | | |



#### 3.0 SYNOPSIS OF STUDY DESIGN

#### 3.1 Purpose of Statistical Analysis Plan

This statistical analysis plan is intended to provide a detailed and comprehensive description of the planned methodology and analysis to be used for the "Automated assessment of pulmonary vein isolation (PVI) using a novel electrophysiology (EP) procedure recording system (CathVision Cube® System)" clinical investigation. This plan is based on the CPVI-002 Clinical Investigation Plan.

#### 3.2 Clinical Investigation Objectives

The main objective in this study is to evaluate the performance of automated PVI Analyzer software with the CathVision Cube® system in radiofrequency (RF), cryo-balloon and pulsed-field ablation (PFA) procedures.

The primary objective of the study is to validate the PVI Analyzer software with a novel EP recording system (CathVision Cube® System) for assisting assessment of isolation status following PVI ablation, while the secondary objectives include the assessment of the accuracy of automated PVI Analyzer classification of pulmonary vein isolation procedures, the determination of the feasibility of "real-time" assessment of PVI analysis, and the assessment of rhythm-dependent performance using the PVI Analyzer and CathVision Cube® System, among other analyses.

### 3.3 Clinical Investigation Design

The PVISION clinical study is a prospective, multi-center study with the CathVision Cube® system and the PVI Analyzer software in pulmonary vein isolation procedures.

The study population is expected to be up to 120 subjects, distributed in three different procedures: RF, cryo-balloon and PFA.

Up to 30 subjects will be enrolled for PFA,

#### 3.4 Endpoints

#### 3.4.1 Primary endpoint

The primary performance endpoint is to validate the PVI Analyzer analysis software with a novel EP recording system (CathVision Cube® System) for assessment of isolation status following PVI ablation. The overall performance of pulmonary vein (PV) isolation classification shall be superior to a specified level of performance.

 Automated PVI Analyzer classification of PV isolation in sinus rhythm (SR) during PVI ablation treatment with a specificity and sensitivity both superior to 80%.



#### 3.4.2 Safety endpoint

The safety endpoint of the Study is to evaluate the adverse events (AEs) and/or device deficiencies reported with the use of the CathVision Cube® System.

it is expected that AEs related to the device

and device deficiencies will be minimal or absent.

#### 3.4.3 Secondary performance endpoints

The secondary performance endpoints have been established to determine the feasibility of time-critical assessment of PVI analysis and rhythm-dependent performance using the PVI Analyzer software with the CathVision Cube® System through the following items:

- Accuracy of automated PVI Analyzer classification of PV isolation in SR during PVI Cryo-balloon ablation
- 2. Accuracy of automated PVI Analyzer classification of PV isolation in SR during RF ablation
- 3. Assessment of automated PVI Analyzer classification of PV isolation in SR after PFA
- 4. Feasibility of continuous "real-time" assessment of isolation
- 5. Feasibility of assessment of isolation during AF rhythm
- Feasibility of assessment of isolation at time of expert-defined isolation before the end of the ablation procedure
- Comparison of device performance on same data recorded by CathVision Cube and Boston Scientific LSPro

#### 3.5 Randomization and blinding

Randomization and blinding are not applicable to this study,

<sup>&</sup>quot;Classification" in secondary performance endpoints also follows the definition described for the primary endpoint.



# 4.0 ANALYSIS CONSIDERATIONS

Enrolled population includes up to 120 patients fulfilling all inclusion criteria,

# 4.1 Analysis Populations

| If any<br>be en | of the exclusion criteria are met, the patient is excluded from the clinical investigation and cannor rolled. |
|---|---|
| 4.1.1 | Intent-to-treat population (ITT) |
| 4.1.2 | Per-protocol treatment (PPT) |
| 4.2 | Data Processing |



#### **Statistical Methods** 4.3

#### **Descriptive statistics for continuous variables**

Continuous variables (e.g., age, beats per minute (BPM), etc.), will be summarized using standard quantitative statistics: number of non-missing observations, mean, standard deviation, median, quartiles and range (minimum and maximum observed values), with 95% confidence intervals (CI) where specified in the table mockups. The number of missing observations, if any, will also be summarized.

#### 4.3.2 Descriptive statistics for categorical variables

For categorical variables (e.g., gender, diabetic status, etc.), results will be summarized using classical frequency statistics: number of non-missing observations and percentages/rates by categories, and where specified in the table mockups, with exact 95% Clopper-Pearson CI.

### 4.4 Endpoint Analysis

| The primary performance endpoint for this investigation is to validate the PVI Analyzer analysis software with a novel EP recording system (CathVision Cube® System) for assessment of isolation status following PVI ablation The performance is evaluated separately for specificity and sensitivity: | 4.4.1 Primary endpoint | |
|---|---|---|
| The performance is evaluated separately for specificity and sensitivity; | software with a novel EP recording system (CathVision Cube® System) for assessment of isola | |
| | The performance is evaluated separately for specificity and sensitivity; | |
| | | 1 |



| a clinically relevant lower limit o |
|---|
| erformance has been established and defined as 80% specificity and 80% sensitivity. |
| 4.2 Safety endpoint |
| he safety endpoint of the study will evaluate the AEs and/or device deficiencies reported with the use |
| the CathVision Cube® System |
| 4.3 Secondary endpoints |
| he secondary performance endpoints will determine the feasibility of time-critical assessment of PV |

The secondary performance endpoints will determine the feasibility of time-critical assessment of PVI analysis and rhythm-dependent performance using the PVI Analyzer software with the CathVision Cube® System.

- Accuracy of automated PVI Analyzer classification of PV isolation in SR during Cryo-balloon ablation.
- Accuracy of automated PVI Analyzer classification of PV isolation in SR during RF ablation.



| • | Assessment of automated PVI Analyzer classification of PV isolation in SR after PFA. |
|---|---|
| | A to see the LDV/LA color and color if the Color of DV/La to Color in NOD |
| • | Automated PVI Analyzer classification of PV isolation in NSR. |
| • | Feasibility of "real-time" assessment of isolation. |
| • | PVI Analyzer classification accuracy at the time of expert-defined isolation. |
| • | Comparison of device performance with conventional system. |
| .5 | Sample Size Calculations |
| | ample size calculation is based on the primary performance endpoint to demonstrate that the PVI |
| | zer software is superior to clinically relevant performance level, as established by prior |
| - | ations. |



| a maximum of 90 subjects will be required. |
|---|
| A cohort of 30 subjects undergoing PFA will be added to the study, and this additional data will be analyzed posteriorly. This PFA cohort does not relate to the primary endpoint and therefore does not affect the primary endpoint analysis nor the sample size calculation. |
| 4.6 |
| 4.7 Timing of Analysis |
| 4.8 Study Success |
| 4.9 |





## 4.10 Handling of Missing Data

Missing data will be counted and summarized in the descriptive analysis for continuous and categorical variables.

Missing data will not be replaced or imputed.

| 4.11 |
|------|
| 4.12 |





#### 5.0 <u>DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA</u>

#### 5.1 Baseline and Demographic Characteristics

The following baseline and demographic variables will be summarized for the subjects enrolled: gender, age, atrial fibrillation and cardiovascular history, cardiac medications, implant procedural characteristics, etc.

#### 5.2 Adverse Events

All of the adverse device effects (ADEs), serious adverse device effects (SADEs), unanticipated adverse device effects (UADEs), and unanticipated serious adverse device effects (USADEs) will be summarized for all subjects who are enrolled in this study,

#### 5.3 Subject Early Termination

Reasons for premature study discontinuation will be collected and summarized when provided or available.

#### 5.4 Protocol Deviation

All protocol deviations, including reasons and associated visit, will be categorized and summarized.

#### 5.5 Number of Subject Imbalance

All efforts will be made to maintain a balanced enrollment among the 4 study centers and among RF and cryo-balloon procedures. A maximum of 25 subjects for RF and 25 subjects for cryo-balloon is set per site. Similarly, balanced enrollment will be attempted for the additional 30 PFA subjects, with a maximum of 15 subjects enrolled per site.



# 6.0 <u>DOCUMENTATION AND OTHER CONSIDERATIONS</u>



## 7.0 APPENDICES

#### **APPENDIX A: MOCK-UP TABLES**

#### Table 1. Subject disposition

| Parameter | Total (N=XX) |
|-------------------|--------------|
| Subjects enrolled | Yes |
| | No |

Abbreviations: n: counts, N: total, %: percentage

Table 2. Study exit

| Parameter | |
|---|---|
| Study exit due to | Study exit due to Completion of study as planned |
| | Discontinued prematurely |
| Reason for withdrawal | Inclusion/exclusion criteria not met |
| | Subject withdrew consent |
| | Subject death |
| | Subject terminated by investigator |
| | Not specified |
| | Other |

Abbreviations: n: counts, N: total, %: percentage

Table 3. Subject enrolment and analysis populations per site

| Site name | Country | Number of subjects<br>enrolled <sup>1</sup> | Number of Screening<br>Failures |
|---|---|---|---|
| Clinique Pasteur Toulouse | France | | |
| UZ Ghent | Belgium | | |
| AZ Sint-Jan Brugge | Belgium | | |
| UZ Brussels | Belgium | | |

<sup>&</sup>lt;sup>1</sup>Values are presented as n/N (%)

Abbreviations: AZ: Algemeen Ziekenhuis; PPT: per-protocol treatment; UZ: Universitair Ziekenhuis.

#### Table 4. Analysis populations

| Site name | PPT population (n/N, %)<br>N=X | ITT population (n/N, %)<br>N=X |
|-----------|--------------------------------|--------------------------------|

Abbreviations: ITT: intent-to-treat; PPT: per-protocol treatment; n: counts, N: total, %: percentage



Table 5. Baseline Demographics, Physical exam, and Vital signs

| Demographics | Total (N=XX) |
|----------------------------------------------|--------------|
| Age, years (at enrolment) <sup>1</sup> | |
| Gender <sup>2</sup> | |
| Female | |
| Male | |
| Height <sup>1</sup> [cm] | |
| Weight <sup>1</sup> [kg] | |
| Systolic Blood Pressure <sup>1</sup> [mmHg] | |
| Diastolic Blood Pressure <sup>1</sup> [mmHg] | |
| Heart Rate <sup>1</sup> [BPM] | |
| Respiratory Rate <sup>1</sup> [breaths/min] | |
| Body Temperature <sup>1</sup> [°C] | |

<sup>1</sup>Values are presented as mean±SD

Abbreviations: BPM: beats per minute; cm: centimetres; ECG: electrocardiogram; kg: kilograms; min: minute; mmHg: millimeter of mercury; n: counts; N: total; SD: standard deviation; °C: degree Celsius; %: percentage

**Table 6. Atrial Fibrillation** 

| Characteristics | Total measurements (N=XX) |
|---------------------------------|---------------------------|
| AF history <sup>1</sup> : | |
| TTM | |
| ECG | |
| Holter | |
| Other | |
| Characteristics | Total Subjects (N=XX) |
| Time from first AF diagnosis to | |
| ablation <sup>2</sup> [days] | |
| AF type <sup>1</sup> : | |
| Paroxysmal | |
| Persistent | |
| Long-term persistent | |

<sup>&</sup>lt;sup>1</sup>Values are presented as n/N (%)

Abbreviations: AF: atrial fibrillation; ECG: electrocardiogram; N: total subjects; TTM: transtelephonic monitor; %: percentage

**Table 7. Cardiovascular History** 

| Characteristics | Total Subjects (N=XX) |
|---|---|
| CHA <sub>2</sub> DS <sub>2</sub> Vasc score <sup>2</sup> | |
| Hypertension <sup>1</sup> : | |
| Yes | |
| No | |
| Structural heart disease1: | |
| Yes | |

<sup>&</sup>lt;sup>2</sup>Values are presented as n/N (%)

<sup>&</sup>lt;sup>2</sup>Values are presented as mean ± SD

<sup>&</sup>lt;sup>3</sup>Values are presented as mean percentage (range) ± SD



| No |
|-------------------------------|
| Diabetes mellitus1: |
| Yes |
| No |
| LVEF <sup>3</sup> |
| LA diameter (mm) <sup>2</sup> |

<sup>&</sup>lt;sup>1</sup>Values are presented as n/N (%)

Abbreviations: CHA₂DS₂Vasc: congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, stroke or transient ischemic attack (TIA), vascular disease, age 65 to 74 years, sex category; LA: left atrial; LVEF: left ventricular ejection fraction; mm: millimeters; N: total subjects; %: percentage

**Table 8. Concomitant medication** 

| Indication | Medication name | n/N (%) |
|------------|-----------------|---------|
| | Any medication | |

Abbreviations: n: counts; N: total; %: percentage

Table 9. Index procedure overview

| Characteristic | Total (N=XX) |
|---|---|
| Procedure type: | |
| Carto RF | |
| Cryoballoon | |
| PFA | |
| General anaesthesia: | |
| Yes | |
| No | |
| Cardioversion performed at the beginning of the procedure: | |
| Yes | |
| No | |
| Patient already in SR | |
| Patient in SR throughout the procedure: | |
| Yes | |
| No | |
| Patient had AF during the procedure and cardioversion was performed: | |
| Yes | |
| No | |
| N/A (patient in SR all the time) | |
| 3D mapping done: | |
| Yes | |
| No | |
| N/A | |

Abbreviations: AF: atrial fibrillation, n: counts; N: total; N/A: not applicable, RF: radiofrequency, SR: sinus rhythm, %: percentage

Table 10. Radiofrequency procedure overview

| Characteristic | Total (N=XX) |
|--------------------------------------------|--------------|
| Name of ablation catheter: "SmartTouch SF" | n/N (%) |
| "SmartTouch" | |
| "Navistar" | |
| <i>u n</i> | |

<sup>&</sup>lt;sup>2</sup>Values are presented as mean ± SD

<sup>&</sup>lt;sup>3</sup>Values are presented as mean percentage (range) ± SD



| Name of circular mapping catheter in the PVs: | n/N (%) |
|---|---|
| "LASSO" | 11/19 (70) |
| "LASSO NAV Eco" | |
| " " | |
| Circular mapping catheter electrodes: | n/N (%) |
| 10 | 11/19 (70) |
| 20 | |
| 20 | |
| Name of CS catheter: | n/N1 (0/ ) |
| Name of CS catheter. | n/N (%) |
| "" | |
| Other setherters | (N.L. (O/) |
| Other catheters: | n/N (%) |
| Yes | |
| No State of the state of the st | (5.1.707.) |
| Data Log Form filled: | n/N (%) |
| Yes | |
| No | |
| Isolation at the right circle after or during deployment of first CLOSE circle: | |
| Yes | |
| At 1-25% circle completion | |
| At 26-50% circle completion | |
| At 51-75% circle completion | |
| At 76-99% circle completion | |
| At 100% circle completion (after full circle) | |
| Carto RF Tag ID | n |
| 3 | Mean |
| | SD |
| | 95% LCLM |
| | 95% UCLM |
| | Q1 |
| | Median |
| | Q3 |
| | Min |
| No find many includes: | Max |
| No first-pass isolation | |
| Additional touch-up ablations | |
| Number of touch-up ablations | n |
| | Mean |
| | SD |
| | 95% LCLM |
| | 95% UCLM |
| | Q1 |
| | Median |
| | Q3 |
| | Min |
| | Max |
| No additional touch-up ablations | |
| Isolation at the left circle after or during deployment of first CLOSE circle: | n/N (%) |
| Yes | '''' |
| At 1-25% circle completion | |
| At 26-50% circle completion | |
| At 51-75% circle completion | |
| At 76-99% circle completion | |
| At 100% circle completion (after full circle) | |
| Corto DE Torr ID | _ |
| Carto RF Tag ID | n |



| | T |
|---|---|
| | Mean |
| | SD |
| | 95% LCLM |
| | 95% UCLM |
| | Q1 |
| | Median |
| | Q3 |
| | Min |
| | Max |
| No first-pass isolation | IVIGA |
| Additional touch-up ablations | |
| | _ |
| Number of touch-up ablations | n<br>Mana |
| | Mean |
| | SD |
| | 95% LCLM |
| | 95% UCLM |
| | Q1 |
| | Median |
| | Q3 |
| | Min |
| | Max |
| No additional touch-up ablations | |
| Pacing to verify isolation at the right circle (after first circle or first circle + | n/N (%) |
| touch ups): | |
| Yes | |
| Correct original isolation assessment | |
| Incorrect original isolation assessment | |
| No | |
| Pacing to verify isolation at the left circle (after first circle or first circle + | n/N (%) |
| touch ups): | |
| Yes | |
| Correct original isolation assessment | |
| Incorrect original isolation assessment | |
| No | |
| 11.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1 | |

Unless otherwise specified, data are presented as n/N (%)

Abbreviations: CS: coronary sinus; ID: identification; LCLM: lower confidence limit for mean; Max: maximum; Min: minimum; n: counts; N: total; PVs: pulmonary veins; Q1: first quartile; Q3: third quartile; RF: radiofrequency; UCLM: upper confidence limit for mean; %: percentage

Table 11. Cryoballoon procedure overview

| Parameter | Total (N=XX) |
|-----------------------------------------------|--------------|
| Name of ablation catheter: | n/N (%) |
| "Arctic Front Advance" | |
| n n | |
| Name of circular mapping catheter in the PVs: | n/N (%) |
| "Achieve" | |
| "Achieve Advance" | |
| Circular mapping catheter electrodes: | n/N (%) |
| 8 | |
| [] | |
| Type of CS catheter: | n/N (%) |
| <i>u n</i> | |
| Other catheters: | n/N (%) |
| Yes | |
| No | |
| Data Log Form filled: | n/N (%) |



| Vac | | |
|---|---|---|
| Yes<br>No | | |
| | RSPV during or after the first freeze attempt: | n/N (%) |
| Yes | There are the mot needed attempt. | 11/14 (70) |
| | After <1 min from start of the freeze | |
| | After <2 min from start of the freeze | |
| | After <3 min from start of the freeze | |
| | After <4 min from start of the freeze | |
| | After 4 min or after session end (waiting time) | |
| No | | |
| | Additional freeze attempts | |
| | 1 | |
| | 2 | |
| | 3 or more | |
| | Isolation achieved | |
| | Isolation not achieved | |
| | No additional freeze attempts | |
| Isolation at the | e RIPV during or after the first freeze attempt: | n/N (%) |
| Yes | | (/0/ |
| | After <1 min from start of the freeze | |
| | After <2 min from start of the freeze | |
| | After <3 min from start of the freeze | |
| | After <4 min from start of the freeze | |
| | After 4 min or after session end (waiting time) | |
| No | | |
| | Additional freeze attempts | |
| | 1 | |
| | 2 | |
| | 3 or more | |
| | Isolation achieved | |
| | Isolation not achieved | |
| | No additional freeze attempts | |
| Isolation at the | LSPV during or after the first freeze attempt: | n/N (%) |
| Yes | | |
| | After <1 min from start of the freeze | |
| | After <2 min from start of the freeze | |
| | After <3 min from start of the freeze | |
| | After <4 min from start of the freeze | |
| No | After 4 min or after session end (waiting time) | |
| No | Additional freeze attempts | |
| | Additional freeze attempts 1 | |
| | 2 | |
| | 3 or more | |
| | Isolation achieved | |
| | Isolation not achieved | |
| | ditional freeze attempts | |
| | e LIPV during or after the first freeze attempt: | n/N (%) |
| Yes | After 44 min from plant of the forces | |
| | After <1 min from start of the freeze | |
| | After <2 min from start of the freeze | |
| | After <3 min from start of the freeze After <4 min from start of the freeze | |
| | After 4 min or after session end (waiting time) | |
| No | And Thin or after session end (waiting time) | |
| 110 | | <u> </u> |



| Additional freeze attempts 1 2 3 or more Isolation achieved Isolation not achieved Isolation not achieved No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation at the LSPV (after all freeze attempts): No N |
|---|
| Isolation achieved Isolation not achieved No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation assessment Incorrect isolation assessment No |
| Isolation achieved Isolation not achieved No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation assessment Incorrect isolation assessment No |
| Isolation achieved Isolation not achieved No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation assessment Incorrect isolation assessment No |
| Isolation not achieved No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No N |
| Isolation not achieved No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No N |
| No additional freeze attempts Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Pacing to verify isolation at the RSPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Incorrect isolation assessment No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| No Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Pacing to verify isolation at the RIPV (after all freeze attempts): Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Yes Correct isolation assessment Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Incorrect isolation assessment No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| No Pacing to verify isolation at the LSPV (after all freeze attempts): n/N (%) |
| Correct isolation assessment |
| Incorrect isolation assessment |
| No |
| Pacing to verify isolation at the LIPV (after all freeze attempts): n/N (%) |
| Yes Yes |
| 1 |
| Correct isolation assessment |
| Incorrect isolation assessment |
| No Unless otherwise specified, data are presented as n/N (%) |

Unless otherwise specified, data are presented as n/N (%)

Abbreviations: CS: coronary sinus; ID: identification; LCLM: lower confidence limit for mean; LIPV: left inferior pulmonary vein; LSPV: left superior pulmonary vein; Max: maximum; Min: minimum; n: counts; N: total; PVs: pulmonary veins; Q1: first quartile; Q3: third quartile; RF: radiofrequency; RIPV: right inferior pulmonary vein; RSPV: right superior pulmonary vein; UCLM: upper confidence limit for mean; %: percentage

Table 12. PFA procedure overview

| Parameter Parame | Total (N=XX) |
|---|---|
| Name of ablation catheter: | n/N (%) |
| u n | |
| Name of circular mapping catheter in the PVs: | n/N (%) |
| "" | (0.1.707.) |
| Number of Circular mapping catheter electrodes: | n/N (%) |
| 8 | |
| Type of CS catheter: | n/N (%) |
| " " | 11/19 (70) |
| Other catheters used: | n/N (%) |
| Yes | 1(75) |
| No | |
| Data Log Form filled: | n/N (%) |
| Yes | |
| No | |
| Isolation at the RSPV after the first PFA attempt: | n/N (%) |
| Yes | |
| No No | |
| Additional freeze attempts | |
| 1 2 | |



| 3 or more | |
|---|---|
| o or more | |
| Isolation achieved | |
| Isolation not achie | |
| No additional freeze attem Isolation at the RIPV after the first PFA att | |
| Yes | empt. 17/14 (70) |
| No | |
| Additional freeze attempts | <b>;</b> |
| 1 | |
| 2 | |
| 3 or more | |
| Isolation achieved | |
| Isolation not achie | |
| No additional freeze attem | npts |
| Isolation at the LSPV after the first PFA at | tempt: n/N (%) |
| Yes | |
| No<br>Additional freeze attempts | , |
| Additional freeze attempts | ' |
| 2 | |
| 3 or more | |
| Isolation achieved | |
| Isolation not achie | eved . |
| No additional freeze attempts Isolation at the LIPV after the first PFA att | empt: n/N (%) |
| Yes | 511pt. 11/14 (76) |
| No | |
| Additional freeze attempts | <b>;</b> |
| 1 | |
| 2 | |
| 3 or more | |
| Isolation achieved | |
| Isolation not achie | |
| No additional freeze attempts | |
| Pacing to verify isolation at the RSPV (after | er all PFA attempts): n/N (%) |
| Yes | _ |
| Correct isolation assessm | |
| Incorrect isolation assessi No | пен |
| Pacing to verify isolation at the RIPV (afte | r all PFA attempts): n/N (%) |
| Yes | (70) |
| Correct isolation assessm | |
| Incorrect isolation assessi | nent |
| No | # DEA (( ) ) |
| Pacing to verify isolation at the LSPV (after | er all PFA attempts): n/N (%) |
| Yes Correct isolation assessm | ent |
| Incorrect isolation assessing | |
| No | |
| Pacing to verify isolation at the LIPV (after | all PFA attempts): n/N (%) |
| Yes | |
| Correct isolation assessm | |
| Incorrect isolation assessi | nent |
| No | |



| Adverse events reported during the procedure | n/N (%) |
|-----------------------------------------------------|---------|
| Yes | |
| No | |
| Protocol deviations identified during the procedure | n/N (%) |
| Yes | . , |
| No | |



Table 13. Overview of PVI Analyzer classification result

| Patient ID | Vein | Label - | PVI Analyzer output* | | Classi | fication result** |
|---|---|---|---|---|---|---|
| | | | Cube | Conventional | Cube | Conventional |
| | LSPV | Baseline | | | | |
| | LSPV | Final | | | | |
| | LIPV | Baseline | | | | |
| | LIPV | Final | | | | |
| | RSPV | Baseline | | | | |
| | RSPV | Final | | | | |
| | RIPV | Baseline | | | | |
| | RIPV | Final | | | | |

<sup>\*</sup>isolated/not isolated

Abbreviations: FN: false negative, FP: false positive, LIPV: left inferior pulmonary vein, LSPV: left superior pulmonary vein, PVI: pulmonary vein isolation, RIPV: right inferior pulmonary vein, RSPV: right superior pulmonary vein, TN: true negative, TP: true positive

Table 14. Patient discharge

| Discharge visit |
|----------------------------------------------|
| Cardiac medications recorded1: |
| Yes |
| No |
| 12 lead ECG performed1: |
| Yes |
| No |
| Systolic Blood Pressure <sup>2</sup> [mmHg] |
| Diastolic Blood Pressure <sup>2</sup> [mmHg] |
| Heart Rate <sup>2</sup> [BPM] |
| Respiratory Rate <sup>2</sup> [breaths/min] |
| Body Temperature <sup>2</sup> [°C] |

<sup>&</sup>lt;sup>1</sup>Values are presented as n/N (%)

Abbreviations: BPM: beats per minute; ECG: electrocardiogram; mmHg: millimetres of mercury; n: counts; N: total; SD: standard deviation; °C: degree Celsius; %: percentage

<sup>\*\*</sup>TN, TP, FN, FP

<sup>&</sup>lt;sup>2</sup>Values are presented as mean±SD



Table 15. Protocol deviations

| Classification | Description | Protocol Deviations<br>(N=XX) (n/N, %) |
|---|---|---|
| Associated visit | Visit 1. Screening | |
| | Visit 2. Procedure | |
| | Visit 3. Discharge | |
| | Not associated to a protocol-defined visit | |
| Type of protocol deviation | Patient consent not obtained or incomplete | |
| | Patient consent not signed & dated by the patient | |
| | Inclusion/exclusion criteria not met | |
| | Required pregnancy test not performed or out of window | |
| | Visit not done | |
| | Assessment not done according to CIP | |
| | Reporting timelines not followed | |
| | Other | |

Abbreviations: CIP: clinical investigation plan; n: counts; N: total; %: percentage

Table 16. Overview of adverse events by severity

| Parameter | | Number of events | Number of subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|---|
| Adverse Event (A | E) reported | | | |
| Severity of AE | Mild | | | |
| | Moderate | | | |
| | Severe | | | |

Abbreviations: AE: adverse event.

Table 17. Adverse events by relation to the study

| Parameter | Relationship | Number of events | Number of subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|---|
| AE relationship to | Device related | | | |
| the study | Procedure related | | | |
| | Other | | | |

Abbreviations: AE: adverse event.

Table 18. Overview of serious adverse events

| Parameter | Number of events | Number of subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|
| Any Serious Adverse Event (SAE) | | | |

Abbreviations: N: total subjects; n: counts



#### **Table 19. Classification of SAEs**

| Classification of SAEs | Number of events | Number of<br>subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|
| Led to death | | | |
| Led to fetal distress, fetal death or a congenital abnormality or birth defect | | | |
| Resulted in a life-threatening illness or injury | | | |
| Resulted in a permanent impairment of a body structure or a body function | | | |
| Resulted in a patient hospitalization or prolonged an existing hospitalization | | | |
| Resulted in a medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function | | | |

Abbreviations: N: total subjects; n: counts

#### Table 20. Overview of serious adverse device effects (SADEs)

| Parameter | Number of events | Number of<br>subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|
| Serious adverse device effect (SADE) incidence | | | |

Abbreviations: N: total subjects; n: counts

#### Table 21. Overview of unanticipated serious adverse device effects (USADEs)

| Parameter | Number of events | Number of<br>subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|
| Serious unanticipated serious adverse device effect (USADE) incidence | | | |

Abbreviations: N: total subjects; n: counts

#### Table 23. Overview of device deficiencies

| Parameter | Number of events | Number of<br>subjects | Rate per subject<br>(n/N, %) N=XX |
|---|---|---|---|
| Device deficiency incidence | | | |

Abbreviations: N: total subjects; n: counts